CLINICAL TRIAL: NCT03940573
Title: A Registry to Further Develop the Understanding of the Real World Use of the Eclipse System for Fecal Incontinence in Women
Brief Title: Pursuit: Real World Use of the Eclipse System
Acronym: PURSUIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pelvalon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA007
Record Dates: First submitted 2019-05-02; First posted 2019-05-07 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): All patients fitted with the device.
  Interventions: Device: Eclipse Insert

INTERVENTIONS:
Device: Eclipse Insert — Rectal Control System.

SUMMARY:
A prospective, open label post-market registry to collect Patient Reported Outcomes and Fitting metrics (e.g. sizes used) in subjects using the Eclipse System in a commercial setting.

DETAILED DESCRIPTION:
Up to 150 subjects enrolled, in up to 25 sites. Population of all adult female patients with Fecal Incontinence (FI) who present at, or are identified at, participating sites are eligible. This includes patients who are newly prescribed Eclipse, and those already using Eclipse who return for an annual renewal visit during the enrollment period.

Includes fitting of the patient for the Eclipse System with collection of relevant health history data. Patients are provided a temporary device for a trial usage period. Multiple device sizes may be attempted to find the correct fit for the patient, at which point the patient is provided with the long term use Eclipse Insert and enters the treatment period.

During the fitting and treatment period, patient experience will be assessed by surveys, St. Mark's (Vaizey) scores, and the validated global PGI-I index (Patient Global Impression of Improvement). Surveys will be perform at the fitting follow up and at 12 months of device usage, and optionally at 3, 6, and 9 months of device usage.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female
2. Diagnosis of Fecal Incontinence
3. Clinician recommendation of the Eclipse System
4. Subject provides informed consent and HIPAA authorization

No Exclusion Criteria.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 150 (Estimated)
Dates: Start 2019-04-19 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Fit Rate | Data collected at fitting visits (max 3 attempts), 5-7 weeks from initial screening
  Proportion of patients successfully fit
Device Size Distribution | Data collected at fitting visits (max 3 attempts), 5-7 weeks from initial screening
  Size distribution of devices among successfully fit patients
St. Mark's Score (Vaizey) | 12 months
  Change from baseline in mean scores (scored 0-24 with 0 = total continence and 24 = total incontinence)
PGI-I Score | 12 months
  Patient global impression of improvement score (7 point scale comparing current condition to baseline, from 1 = very much better to 7 = very much worse)

SECONDARY OUTCOMES:
St. Mark's Score (Vaizey) | 3 months
  Change from baseline in mean scores (scored 0-24 with 0 = total continence and 24 = total incontinence)
St. Mark's Score (Vaizey) | 6 months
  Change from baseline in mean scores (scored 0-24 with 0 = total continence and 24 = total incontinence)
St. Mark's Score (Vaizey) | 9 months
  Change from baseline in mean scores (scored 0-24 with 0 = total continence and 24 = total incontinence)
PGI-I Score | 3 months
  Patient global impression of improvement score (7 point scale comparing current condition to baseline, from 1 = very much better to 7 = very much worse)
PGI-I Score | 6 months
  Patient global impression of improvement score (7 point scale comparing current condition to baseline, from 1 = very much better to 7 = very much worse)e
PGI-I Score | 9 months
  Patient global impression of improvement score (7 point scale comparing current condition to baseline, from 1 = very much better to 7 = very much worse)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pettit, MD, Principal Investigator — Mayo Clinic
Locations (6):
- United States (6):
  - The American Association of Female Pelvic Medicine, Agoura Hills, California
  - The Ob-Gyn and Incontinence Center, Arcadia, California
  - Long Beach Urogynecology, Long Beach, California
  - Florida Urogynecology, LLC, Jacksonville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Princeton Urogynecology, Princeton, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pelvalon, Eclipse manufacturer and Study Sponsor, website — http://eclipsesystem.com/

DOCUMENTS (1):
  • Study Protocol (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT03940573/Prot_000.pdf